CLINICAL TRIAL: NCT02227901
Title: Phase I Trial of R115777 With Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Tipifarnib, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01809; NCI-2014-01809 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-03-C-0189; NABTC-0202; NABTC02-02 (Other: Adult Brain Tumor Consortium); NABTC-02-02 (Other: CTEP); U01CA062399 (NIH)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-09

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — tipifarnib; Temozolomide

ARMS (1):
- Treatment (tipifarnib, EBRT, temozolomide) (Experimental): TIPIFARNIB: Patients receive tipifarnib PO BID on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  CONCURRENT CHEMOTHERAPY DURING RADIATION THERAPY: Within 5-9 days after starting tipifarnib, patients undergo EBRT daily and receive temozolomide PO daily for 6 weeks.
  POST-RADIATION CHEMOTHERAPY: Beginning at week 10 post-radiation therapy, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for 1 year or 12 complete courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tipifarnib; Radiation: External Beam Radiation Therapy; Drug: Temozolomide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT
Drug: Temozolomide — Given PO
  Other Names: TMZ
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of tipifarnib when given together with radiation therapy and temozolomide in treating patients with newly diagnosed glioblastoma multiforme. Tipifarnib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving tipifarnib together with radiation therapy and temozolomide may be a better way to treat glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish maximum tolerated dose (MTD) for tipifarnib (R115777) in combination with temozolomide with radiation in patients not on enzyme-inducing anti-epileptic drugs (EIAEDs).

II. To define the safety of R115777 in combination with temozolomide with radiation in this patient population.

III. To assess for evidence of antitumor activity in this patient population.

OUTLINE: This is a dose-escalation study of tipifarnib.

TIPIFARNIB: Patients receive tipifarnib orally (PO) twice daily (BID) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

CONCURRENT CHEMOTHERAPY DURING RADIATION THERAPY: Within 5-9 days after starting tipifarnib, patients undergo external beam radiation therapy (EBRT) daily and receive temozolomide PO daily for 6 weeks.

POST-RADIATION CHEMOTHERAPY: Beginning at week 10 post-radiation therapy, patients receive temozolomide PO on days 1-5. Treatment repeats every 28 days for 1 year or 12 complete courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have histologically proven intracranial glioblastoma multiforme (GBM) or gliosarcoma (GS)
* Diagnosis will have been established by biopsy or resection within 4 weeks prior to registration
* Patients must not have received previous radiotherapy to the brain
* Patients must not have received cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy directed against the brain tumor; patients who received Gliadel wafers will be excluded; patients may have received or be receiving corticosteroids, non-EIAEDs, analgesics, and other drugs to treat symptoms or prevent complications
* Cranial magnetic resonance imaging (MRI) or contrast computed tomography (CT) must have been performed within 21days of study entry; the use of MRI rather than CT is preferred; the same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement; if the surgical procedure was a resection, cranial MRI or contrast CT performed with 96 hours of resection is preferred but not required; patients without measurable or assessable disease are eligible
* Patients must have a plan to begin partial brain radiotherapy within 5-9 days after beginning R115777, and within 35 days (5 weeks) of the surgical procedure that established the diagnosis; radiotherapy must be given at the Radiation Oncology Department of the registering Adult Brain Tumor Consortium (ABTC) institution; radiotherapy must be given by external beam to a partial brain field in daily fractions of 2.0 Gray (Gy), to a planned total dose to the tumor of 60.0 Gy; stereotactic radiosurgery and brachytherapy will not be allowed
* Patients must be willing to forego other drug therapy against the tumor while being treated with R115777 and temozolomide
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must sign an authorization for the release of their protected health information; patients must be registered with the Adult Brain Tumor Consortium Central Office (ABTC CO) prior to treatment with study drug
* A life expectancy > 8 weeks
* Patients must have a Karnofsky performance status of >= 60
* White blood cells (WBC) >= 3,000/ul
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3
* Hemoglobin >= 10 gm/dl
* Bone marrow function tests must be performed within 14 days prior to registration
* Eligibility level for hemoglobin may be reached by transfusion
* Serum glutamic oxaloacetic transaminase (SGOT) < 2 times upper limit of normal (ULN) and the test must be performed within 14 days prior to registration; if above the institutional upper limit of normal but < 2 times institutional upper limit of normal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient
* Bilirubin < 2 times ULN and the test must be performed within 14 days prior to registration; if above the institutional upper limit of normal but < 2 times institutional upper limit of normal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient
* Creatinine < 1.5 mg/dL before starting therapy and the test must be performed within 14 days prior to registration
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy; patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* No exclusion to this study will be based on race; minorities will actively be recruited to participate
* Patients must not have active infection
* Women must not be pregnant or breast-feeding, and women with reproductive potential must practice adequate contraception
* Patients must not be on chronic Coumadin therapy for prior medical problems (e.g. cardiac valve prophylaxis); this is due to a presumed interaction with Coumadin and ZARNESTRA leading to a significant increase in international normalized ratio (INR); patients who develop or have recently developed a deep venous thrombosis or pulmonary embolism who are on or will take Coumadin will be allowed to participate; however, the investigator should be prepared to monitor patients INR closely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-09; Primary Completion 2007-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of tipifarnib, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 | At week 10
  Safety variables will be summarized by descriptive statistics.
MTD of tipifarnib, defined as the dose level at which 0 or 1/6 patients experience DLT with the next higher dose having at least 2/3 or 2/6 patients encountering DLT, graded according to the NCI CTCAE v4.0 | Up to week 10
  Safety variables will be summarized by descriptive statistics.

SECONDARY OUTCOMES:
Incidence of adverse events of tipifarnib in combination with EBRT and temozolomide, graded according to the NCI CTCAE v4.0 | Up to 5 years
  Safety variables will be summarized by descriptive statistics. Adverse events that occur will be reported for each dose level and described in terms of incidence and severity. Parameters will be described based on the CTCAE severity grading. Distribution by CTCAE severity grade (when applicable) and clinical relevance will be given.
Anti-tumor activity of tipifarnib | Up to 5 years
  A descriptive analysis of evidence of antitumor activity will be provided based on clinical, radiographic, and biologic assessments of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Cloughesy, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States